CLINICAL TRIAL: NCT06855381
Title: Ultrasound-guided Interscalene Brachial Plexus Block: Single Bolus Injection Versus Continuous Catheter Placement in Arthroscopic Rotator Cuff Repair-a Prospective Randomized Unblinded Trial
Brief Title: Ultrasound-guided Interscalene Brachial Plexus Block: Single Bolus Vs Continuous Catheter Placement in Arthroscopic Rotator Cuff Repair
Acronym: ISB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, Doctor, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: unifg
Record Dates: First submitted 2025-02-07; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Anesthesia
Keywords: interscalene block, pain management, regional anesthesia, shoulder arthroscopy
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- effectiveness of interscalene brachial plexus single-shot (Active Comparator): An ultrasound-guided peripheral nerve block puncture will be performed from the lateral to the medial side of the neck. In this group a 22G 50 mm needle will be used
  Interventions: Procedure: single bolus injection
- continuous interscalene brachial plexus block (Experimental): An ultrasound-guided peripheral nerve block puncture will be performed from the lateral to the medial side of the neck. In this arm, a 22G 50 mm SonoPlex needle with an indwelling cannula will be used.
  Interventions: Procedure: the ISBC group, SonoPlex needle and E-catheter

INTERVENTIONS:
Procedure: the ISBC group, SonoPlex needle and E-catheter — in the ISBC group, a 22G 50 mm SonoPlex needle with an indwelling cannula will be used. The E-catheter will be inserted into the indwelling cannula.
  Arms: continuous interscalene brachial plexus block
Procedure: single bolus injection — An ultrasound-guided peripheral nerve block puncture will be performed from the lateral to the medial side of the neck. In this group a 22G 50 mm needle will be used
  Arms: effectiveness of interscalene brachial plexus single-shot

SUMMARY:
Shoulder arthroscopy is a minimally invasive procedure frequently used for rotator cuff repair. Patients may experience severe postoperative (PO) pain, that can last for a month and can influence successful rehabilitation. Our study aimes to evaluate the effectiveness of interscalene brachial plexus single-shot (ISBSS) versus continuous interscalene brachial plexus block (ISBC) in controlling perioperative pain and avoiding PO pain chronicization. This prospective randomized unblinded trial hypothesizes that the PO perineuronal infusion using a continuous ambulatory delivery device pump gives better pain control and outcomes than ISBSS during the long-term follow-up period.

DETAILED DESCRIPTION:
Blocks will be performed under ultrasound guidance with 15 - 20 mL of 0.75 % ropivacaine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia (ASA) physical status of 1 to 2,
* Body Mass Index (BMI) of less than 30 kg/m²,
* paitents undergoing shoulder arthroscopy for small to medium rotator cuff tears.

Exclusion Criteria:

* skin infection on the puncture site,
* coagulopathy
* brachial plexus neuropathy
* alcohol or drug abuse
* diabetes
* severe lung disease
* history of allergy to one or more study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 24 hour, 48 hour, 72 hour, 7 day
  Tha pain severity will be evaluated by NRS scale

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico, Foggia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uno T, Mura N, Yuki I, Oishi R, Takagi M. The effect of continuous interscalene brachial plexus block for arthroscopic rotator cuff repair. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2024 Feb 2;36:6-12. doi: 10.1016/j.asmart.2024.01.004. eCollection 2024 Apr. PMID 38344106
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10850117/